CLINICAL TRIAL: NCT04346628
Title: A Phase 2 Randomized, Double Blinded, Placebo Controlled Study of Oral Favipiravir Compared to Standard Supportive Care in Subjects With Mild or Asymptomatic COVID-19
Brief Title: Oral Favipiravir Compared to Placebo in Subjects With Mild COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56032
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Results first posted 2022-04-21 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Sars-CoV2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Favipiravir (Experimental): In addition to SOC, participants will receive favipiravir for 10 days, and be evaluated for health outcomes through day 28.
  Interventions: Drug: Favipiravir; Other: Standard of care treatment
- Placebo (Active Comparator): In addition to SOC, participants will receive placebo to match favipiravir for 10 days, and be evaluated for health outcomes through day 28.
  Interventions: Drug: Placebo; Other: Standard of care treatment

INTERVENTIONS:
Drug: Favipiravir — Favipiravir administered orally, 1800 mg on the first dose (day 1) followed by 800 mg twice daily for the next 9 days (days 2-10).
  Arms: Favipiravir
Drug: Placebo — Placebo to match favipiravir administered orally through day 10.
  Arms: Placebo
Other: Standard of care treatment — Standard of care treatment for COVID-19 infection

SUMMARY:
The objective of this study is to evaluate the efficacy of oral favipiravir plus standard of care treatment (SOC) compared with placebo plus SOC in reducing the duration of shedding of SARS-CoV2 virus in patients with mild or asymptomatic COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 disease:

  * If symptomatic, presence of mild to moderate symptoms without signs of respiratory distress, with positive for SARS-CoV-2 diagnostic assay within 72 hours prior to.informed consent.
  * If asymptomatic, initial diagnosis obtained no more than 72 hours prior to informed consent
* Subject agrees to maintain home or other quarantine as recommended by the study physician, except to visit the study site as required by the protocol
* Members of the same household may participate in the study as long as the inclusion and exclusion criteria are met
* Males must be sterile, OR agree not to donate semen AND agree to strictly adhere to contraceptive measures during the study and for seven days following the last dose of study medication
* Females must be unable to bear children, OR ensure that their male partner is incapable of fathering a child, OR, if of childbearing potential will strictly adhere to contraceptive measures during the study and for seven days following the last dose of study medication
* Females must agree to stop breast-feeding prior to first dose of study drug and through seven days after completing therapy
* Females must have a negative pregnancy test at screening
* Participant agrees to maintain home or other quarantine as recommended by the study physician, except to visit the study site as required by the protocol

Exclusion Criteria:

* Concomitant bacterial respiratory infection documented by respiratory culture. NOTE: Subjects on empirical antibiotic treatment for possible but unproven bacterial pneumonia, but who are positive for SARS-CoV-2, are allowed in the study (will be randomized to the same treatment to maintain blinding).
* History of abnormal uric acid metabolism.
* History of hypersensitivity to an anti-viral nucleoside-analog drug targeting a viral RNA polymerase.
* Abnormal laboratory test results at screening:
* Use of adrenocorticosteroids (except topical or inhaled preparations or oral preparations equivalent to or less than 10 mg of oral prednisone) or immunosuppressive or immunomodulatory drugs (e.g., immunosuppressants, anticancer drugs, interleukins, interleukin antagonists or interleukin receptor blockers). NOTE: Treatment of study participants following institutional COVID-19 treatment policies or guidelines, including the use of immunomodulatory medications, is permitted. This excludes treatment with agents that have the potential for direct antiviral activity, including convalescent plasma and NO, and co-enrollment into other clinical studies that evaluate investigational agents for COVID-19.
* Serious chronic disease (e.g., human immunodeficiency virus [HIV], cancer requiring chemotherapy within the preceding 6 months, and/or moderate or severe hepatic insufficiency).
* Previously received favipiravir within the past 30 days.
* Advanced kidney disease
* Advanced liver disease
* History of alcohol or drug abuse in the previous two years.
* Psychiatric illness that is not well controlled (defined as stable on a regimen for more than one year).
* Taken another investigational drug within the past 30 days.
* Seemed by the Investigator to be ineligible for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne (Bonnie) A Maldonado, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share individual participant data (IPD).

REFERENCES:
- [Result] Holubar M, Subramanian A, Purington N, Hedlin H, Bunning B, Walter KS, Bonilla H, Boumis A, Chen M, Clinton K, Dewhurst L, Epstein C, Jagannathan P, Kaszynski RH, Panu L, Parsonnet J, Ponder EL, Quintero O, Sefton E, Singh U, Soberanis L, Truong H, Andrews JR, Desai M, Khosla C, Maldonado Y. Favipiravir for Treatment of Outpatients With Asymptomatic or Uncomplicated Coronavirus Disease 2019: A Double-Blind, Randomized, Placebo-Controlled, Phase 2 Trial. Clin Infect Dis. 2022 Nov 30;75(11):1883-1892. doi: 10.1093/cid/ciac312. PMID 35446944
- [Derived] Jacobson KB, Rao M, Bonilla H, Subramanian A, Hack I, Madrigal M, Singh U, Jagannathan P, Grant P. Patients With Uncomplicated Coronavirus Disease 2019 (COVID-19) Have Long-Term Persistent Symptoms and Functional Impairment Similar to Patients with Severe COVID-19: A Cautionary Tale During a Global Pandemic. Clin Infect Dis. 2021 Aug 2;73(3):e826-e829. doi: 10.1093/cid/ciab103. PMID 33624010

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 385 participants were assessed for eligibility; 149 participants were enrolled and randomized.
Groups:
- Placebo: In addition to standard of care (SOC) treatment for COVID-19 infection, participants were randomized to receive placebo to match favipiravir for 10 days, and to be evaluated for health outcomes through day 28.
- Favipiravir: In addition to SOC treatment for COVID-19 infection, participants were randomized to receive favipiravir for 10 days, and to be evaluated for health outcomes through day 28. Favipiravir was administered orally, 1800 mg on the first dose (day 1) followed by 800 mg twice daily for the next 9 days (days 2-10).
Period: Overall Study
Arm/Group | Placebo | Favipiravir
Started | 74 | 75
Intention-to-treat (ITT) Analysis Set | 74 | 75
Symptomatic Modified ITT (smITT) Analysis Set (Participant reported at least one symptom other than mild cough, mild fatigue, or decreased taste/smell at baseline.) | 70 | 65
Modified ITT (mITT) Analysis (Participant was symptomatic with positive RT-PCR result at baseline.) | 57 | 59
Completed | 68 | 62
Not Completed | 6 | 13
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrew (had personal reasons) | 2 | 5
Not completed — Withdrew (medication intolerant) | 0 | 3
Not completed — Withdrew (declined intervention) | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed for the symptomatic modified ITT (smITT) Analysis Set (participants who reported at least one symptom other than mild cough, mild fatigue, or decreased taste/smell at baseline), and for the modified ITT (mITT) Analysis Set (participants who were symptomatic with positive RT-PCR result at baseline).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Favipiravir | Total
Number analyzed (Participants) | 70 | 65 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  years
    smITT analysis set | 42.8 (12.6) | 42.5 (12.0) | 42.6 (12.3)
    mITT analysis set: number analyzed (Participants) | 57 | 59 | 116
    mITT analysis set | 43.4 (12.8) | 42.9 (12.3) | 43.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  Participants
    smITT Analysis Set: Female | 37 | 32 | 69
    smITT Analysis Set: Male | 33 | 33 | 66
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set: Female | 29 | 28 | 57
    mITT Analysis Set: Male | 28 | 31 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  Participants
    Latinx - smITT Analysis Set | 29 | 28 | 57
    Latinx - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    Latinx - mITT Analysis Set | 24 | 26 | 50
    White - smITT Analysis Set | 26 | 22 | 48
    White - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    White - mITT Analysis Set | 21 | 19 | 40
    Asian - smITT Analysis Set | 7 | 6 | 13
    Asian - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    Asian - mITT Analysis Set | 5 | 6 | 11
    Native Hawaiian/ Pacific Islander - smITT Analysis Set | 1 | 3 | 4
    Native Hawaiian/ Pacific Islander - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    Native Hawaiian/ Pacific Islander - mITT Analysis Set | 1 | 2 | 3
    Other/Unknown - smITT Analysis Set | 7 | 6 | 13
    Other/Unknown - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    Other/Unknown - mITT Analysis Set | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants] — Participants in the smITT Analysis Set.
  Participants
    United States | 70 | 65 | 135
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  kg/m^2
    smITT Analysis Set | 28.9 (5.9) | 28.0 (5.8) | 28.4 (5.8)
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 29.3 (6.0) | 27.8 (5.7) | 28.5 (5.9)
Comorbid Conditions [Count of Participants; unit: Participants] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set with available data.
  Participants
    None - smITT Analysis Set: number analyzed (Participants) | 63 | 63 | 126
    None - smITT Analysis Set | 48 | 47 | 95
    None - mITT Analysis Set: number analyzed (Participants) | 50 | 55 | 105
    None - mITT Analysis Set | 39 | 41 | 80
    Diabetes mellitus - smITT Analysis Set: number analyzed (Participants) | 63 | 63 | 126
    Diabetes mellitus - smITT Analysis Set | 4 | 8 | 12
    Diabetes mellitus - mITT Analysis Set: number analyzed (Participants) | 50 | 55 | 105
    Diabetes mellitus - mITT Analysis Set | 3 | 7 | 10
    Hypertension - smITT Analysis Set: number analyzed (Participants) | 63 | 63 | 126
    Hypertension - smITT Analysis Set | 8 | 6 | 14
    Hypertension - mITT Analysis Set: number analyzed (Participants) | 50 | 55 | 105
    Hypertension - mITT Analysis Set | 5 | 5 | 10
    Chronic lung disease - smITT Analysis Set: number analyzed (Participants) | 63 | 63 | 126
    Chronic lung disease - smITT Analysis Set | 3 | 2 | 5
    Chronic lung disease - mITT Analysis Set: number analyzed (Participants) | 50 | 55 | 105
    Chronic lung disease - mITT Analysis Set | 3 | 2 | 5
Asymptomatic [Count of Participants; unit: Participants] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  Participants
    smITT Analysis Set | 0 | 0 | 0
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 1 | 3 | 4
Days from symptom onset to randomization [Median (Inter-Quartile Range); unit: days] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  days
    smITT Analysis Set | 5 [4 to 7] | 5 [3 to 7] | 5 [4 to 7]
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 5 [4 to 6] | 5 [3 to 7] | 5 [4 to 7]
Number of symptoms reported at randomization [Median (Inter-Quartile Range); unit: symptoms] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  symptoms
    smITT Analysis Set | 6 [4 to 9] | 6 [4 to 8] | 6 [4 to 9]
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 6 [4 to 9] | 6 [4 to 8.5] | 6 [4 to 9]
Symptoms at randomization [Count of Participants; unit: Participants] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  Participants
    Fever - smITT Analysis Set | 3 | 1 | 4
    Fever - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    Fever - mITT Analysis Set | 2 | 1 | 3
    Cough/dyspnea - smITT Analysis Set | 48 | 47 | 95
    Cough/dyspnea - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    Cough/dyspnea - mITT Analysis Set | 44 | 42 | 86
    Fatigue - smITT Analysis Set | 51 | 47 | 98
    Fatigue - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    Fatigue - mITT Analysis Set | 41 | 40 | 81
    Joint pain - smITT Analysis Set | 20 | 22 | 42
    Joint pain - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    Joint pain - mITT Analysis Set | 18 | 20 | 38
    Myalgias - smITT Analysis Set | 42 | 38 | 80
    Myalgias - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    Myalgias - mITT Analysis Set | 36 | 36 | 72
    Headache - smITT Analysis Set | 45 | 43 | 88
    Headache - mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    Headache - mITT Analysis Set | 37 | 40 | 77
Received at least one dose of COVID-19 vaccine [Count of Participants; unit: Participants] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  Participants
    smITT Analysis Set | 2 | 0 | 2
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 2 | 0 | 2
Seropositive [Count of Participants; unit: Participants] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  Participants
    smITT Analysis Set | 11 | 9 | 20
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 4 | 6 | 10
Anterior nares RT-PCR Ct [Median (Inter-Quartile Range); unit: cycles] — Cycle threshold (Ct) denotes how many PCR cycles are required before the SARS-CoV-2 viral RNA reached a detectable level. Higher Ct values correspond to lower viral copy numbers. For reference, Ct values of 20 correspond to ~2.12 x 106 viral copies per milliliter, while a Ct value of 40 is undetectable and is considered the lower limit of detection of this RT-PCR test for SARS-CoV-2. RT-PCR: reverse transcription-polymerase chain reaction. Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  cycles
    smITT Analysis Set | 28.3 [23.2 to 38.4] | 24.3 [20.7 to 31.9] | 26.2 [21.6 to 34.2]
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 25.1 [22.2 to 28.9] | 22.2 [19.7 to 27.2] | 24.0 [21.0 to 27.8]
Oropharyngeal RT-PCR positivity [Count of Participants; unit: Participants] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  Participants
    smITT Analysis Set | 52 | 53 | 105
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 50 | 54 | 104
Aspartate aminotransferase (AST) [Median (Inter-Quartile Range); unit: units/L] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  units/L
    smITT Analysis Set | 29.5 [25.8 to 39.3] | 29.0 [25.0 to 34.0] | 29.0 [25.0 to 36.0]
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 32.0 [26.0 to 42.5] | 29.0 [25.0 to 34.0] | 29.0 [25.0 to 36.8]
Alanine Aminotransferase (ALT) [Median (Inter-Quartile Range); unit: units/L] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  units/L
    smITT Analysis Set | 24.5 [18.8 to 46.5] | 25.0 [19.0 to 37.0] | 25.0 [19.0 to 40.0]
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 29.0 [20.0 to 48.0] | 25.0 [19.5 to 38.0] | 25.5 [20.0 to 40.8]
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  mg/dL
    smITT Analysis Set | 0.8 [0.7 to 1.0] | 0.8 [0.6 to 1.0] | 0.8 [0.64 to 1.0]
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 0.8 [0.6 to 1.0] | 0.8 [0.6 to 1.0] | 0.8 [0.61 to 1.0]
Uric acid [Median (Inter-Quartile Range); unit: mg/dL] — Population: Participants in the smITT Analysis Set and the mITT Analysis Set.
  mg/dL
    smITT Analysis Set | 4.5 [3.5 to 5.6] | 4.4 [3.9 to 5.3] | 4.5 [3.6 to 5.35]
    mITT Analysis Set: number analyzed (Participants) | 57 | 59 | 116
    mITT Analysis Set | 4.5 [3.5 to 5.8] | 4.4 [3.9 to 5.3] | 4.5 [3.7 to 5.5]

OUTCOME MEASURES:

1. Primary Outcome: Time Until Cessation of Oral Shedding of SARS-CoV-2 Virus
Description: Time in days from randomization to the first two negative results of nasal and/or oropharyngeal swab.
Time Frame: Up to 28 days
Population: Modified intention-to-treat (mITT) Analysis Set (participants who were symptomatic with positive RT-PCR result at baseline)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Favipiravir
Number analyzed (Participants) | 57 | 59
days | 13 [9 to 14] | 14 [9 to 21]
Statistical Analysis 1: Comparison: Placebo vs Favipiravir; Test type: Superiority; p = 0.24, Cox proportional hazards model — The final test was performed at the alpha = 0.04999 level of significance, adjusted for age group and sex; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.48 to 1.20] — Hazard ratio adjusted for age and sex

2. Secondary Outcome: Sars-CoV-2 Viral Load
Description: Viral load (nucleic acid) will be assessed by RT-PCR Ct over time. Cycle threshold (Ct) denotes how many PCR cycles are required before the SARS-CoV-2 viral RNA reached a detectable level. Higher Ct values correspond to lower viral copy numbers. For reference, Ct values of 20 correspond to ~2.12 x 106 viral copies per milliliter, while a Ct value of 40 is undetectable and is considered the lower limit of detection of this RT-PCR test for SARS-CoV-2.
Time Frame: Up to 28 days
Population: mITT Analysis Set (participants who were symptomatic with positive RT-PCR result at baseline)
Measure: Median (Inter-Quartile Range); unit: cycles
Arm/Group | Placebo | Favipiravir
Number analyzed (Participants) | 57 | 59
cycles
  Day 1 | 25.1 [22.2 to 28.9] | 22.2 [19.7 to 27.2]
  Day 5 | 27.3 [25.2 to 33.5] | 27.9 [24.7 to 31.9]
  Day 10 | 37.3 [33.1 to 40.0] | 40.0 [33.1 to 40.0]
  Day 28 | 40.0 [40.0 to 40.0] | 40.0 [40.0 to 40.0]

3. Secondary Outcome: Count of Participants With Clinical Worsening of COVID-19 Disease
Description: Clinical worsening is reported as the number of participants with hospitalization or emergency department (ED) visits.
Time Frame: Up to 28 days
Population: Intention-to-treat (ITT) analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Favipiravir
Number analyzed (Participants) | 74 | 75
Participants
  Hospitalization | 4 | 0
  ED visit | 7 | 5
Statistical Analysis 1: Comparison: Placebo vs Favipiravir; Difference in hospitalizations; Test type: Superiority; p = 0.06, Fisher Exact — A p-value of 0.05 would have been considered statistically significant
Statistical Analysis 2: Comparison: Placebo vs Favipiravir; Difference in ED visits; Test type: Superiority; p = 0.56, Fisher Exact — A p-value of 0.05 would have been considered statistically significant

4. Secondary Outcome: Count of Participants With Development of SARS-CoV-2 Antibodies
Time Frame: Up to 28 days
Population: ITT analysis set; participants with available data at each time point are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Favipiravir
Number analyzed (Participants) | 74 | 75
Participants
  Baseline: number analyzed (Participants) | 63 | 65
  Baseline | 12 | 9
  Day 28: number analyzed (Participants) | 55 | 50
  Day 28 | 47 | 40

5. Secondary Outcome: Time Until Cessation of Symptoms
Description: Time until cessation of symptoms is reported as days until initial resolution and sustained resolution of symptoms.
Time Frame: Up to 28 days
Population: Symptomatic Modified Intention-to-treat (smITT) Analysis Set (participants reported at least one symptom other than mild cough, mild fatigue, or decreased taste/smell at baseline)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Favipiravir
Number analyzed (Participants) | 70 | 65
days
  Initial resolution of symptoms | 14 [11 to 18] | 15 [12 to 26]
  Sustained resolution of symptoms | 24 [21 to NA] — Not estimable (curve did not reach the 75th percentile) | NA [26 to NA] — Not estimable (curve did not reach either the median or the 75th percentile)
Statistical Analysis 1: Comparison: Placebo vs Favipiravir; Difference in days until initial resolution of symptoms; Test type: Superiority; p = 0.43, Cox proportional hazards model — A p-value of 0.05 would have been considered statistically significant; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.54 to 1.29] — Hazard ratio adjusted for age and sex
Statistical Analysis 2: Comparison: Placebo vs Favipiravir; Difference in days until sustained resolution of symptoms; Test type: Superiority; p = 0.59, Cox proportional hazards model — A p-value of 0.05 would have been considered statistically significant; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.52 to 1.45] — Hazard ratio adjusted for age and sex

6. Secondary Outcome: Count of Participant With Absence of Development of Any Symptoms
Description: This outcome will be assessed in patient who are asymptomatic of COVID-19 infection at the time of enrollment
Time Frame: Up to 28 days
Population: smITT Analysis Set (participants reported at least one symptom other than mild cough, mild fatigue, or decreased taste/smell at baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Favipiravir
Number analyzed (Participants) | 70 | 65
Participants | 2 | 5

7. Secondary Outcome: Cmax of Favipiravir
Description: Cmax is a pharmacokinetic parameter that measures the maximum concentration of drug in plasma.
Time Frame: Days 1 and 10 (samples taken 30 minutes prior to and 1 hour following favipiravir administration)
Population: Data were not collected for this outcome measure.
Arm/Group | Placebo | Favipiravir
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Cmin of Favipiravir
Description: Cmin is a pharmacokinetic parameter that measures the minimum concentration of drug in plasma.
Time Frame: Days 1 and 10 (samples taken 30 minutes prior to and 1 hour following favipiravir administration)
Population: Data were not collected for this outcome measure.
Arm/Group | Placebo | Favipiravir
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Placebo | Favipiravir
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 1/74 | 0/75
Other Adverse Events (participants affected / at risk) | 0/74 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | Favipiravir (N=75)
Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT04346628/Prot_SAP_000.pdf